CLINICAL TRIAL: NCT07263425
Title: Efficacy and Safety of Intrathecal Administration of Thiotepa in Combination With Trastuzumab Via the Ommaya Reservoir in Breast Cancer With Leptomeningeal Metastasis: a Phase II Multicenter Clinical Trial
Brief Title: Efficacy and Safety of Intrathecal Administration of Thiotepa in Combination With Trastuzumab in Breast Cancer With Leptomeningeal Metastasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: The Affiliated Brain Hospital of Nanjing Medical University (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ommaya 02
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Leptomeningeal Metastasis of HER2-positive Breast Cancer
Keywords: Trastuzumab; Thiotepa; intrathecal chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Intrathecal chemotherapy group Patients received intrathecal 150mg Trastuzumab combination with 10mg thiotepa once every three weeks until an event that meets the criteria for termination occurs.
  Interventions: Drug: Intrathecal Administration of Thiotepa in Combination with Trastuzumab via the Ommaya Reservoir

INTERVENTIONS:
Drug: Intrathecal Administration of Thiotepa in Combination with Trastuzumab via the Ommaya Reservoir — Intrathecal chemotherapy group Patients received intrathecal 150mg Trastuzumab combination with 10mg thiotepa once every three weeks until an event that meets the criteria for termination occurs.

SUMMARY:
Evaluate the efficacy and safety of Intrathecal Administration of Thiotepa in Combination with Trastuzumab via the Ommaya Reservoir in Breast Cancer with Leptomeningeal Metastasis

DETAILED DESCRIPTION:
This was a II, single-arm, prospective, multicenter study designed to estimate the efficacy and safety of intrathecal administration of thiotepa in combination with Trastuzumab via the Ommaya Reservoir in HER2-positive breast cancer with leptomeningeal metastasis.

The primary end point was iORR [complete response (CR) + partial response (PR)] according to RANO-LM. Scoring based on radiographic assessment in leptomeningeal metastases . A composite score (total score) is calculated and compared with the baseline total score. A 25% worsening in the current score relative to baseline defines radiographic progressive disease. A 50% improvement in the current score defines a radiographic partial response. Resolution of all baseline radiographic abnormalities defines a complete response. All other situations define stable disease. The secondary end points were changes in iPFS,PFS, OS, and exploratory analysis of the relationship between molecular markers and therapeutic efficacy.

This study is planned to include 26 patients with leptomeningeal metastasis from breast cancer who meet the entry criteria.

ELIGIBILITY:
Inclusion Criteria:The subjects must meet all of the following criteria simultaneously:

* Histologically or cytologically confirmed HER-2 positive breast cancer (immunohistochemistry indicates HER-2 3+ and/or fluorescence in situ hybridization indicates HER-2 gene amplification)
* Diagnosed with breast cancer with leptomeningeal metastasis based on cerebrospinal fluid cytology combined with central nervous system function and brain imaging findings
* The patient has an Ommaya reservoir implanted or is eligible for implantation
* KPS ≥ 30
* Adequate bone marrow and liver and kidney function reserves: absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, hemoglobin ≥ 90 g/L. International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 x ULN. Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN. Total serum bilirubin ≤ 1.5 x ULN (patients with Gilbert's syndrome can be enrolled if total bilirubin < 3 x ULN). Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN; if the patient has liver metastasis, this criterion is AST and ALT ≤ 5 x ULN.
* Female, aged between 18 and 75 years old
* Left ventricular ejection fraction (LVEF) > 50%
* Voluntary signing of informed consent form

Exclusion Criteria:

Patients meeting any of the following criteria are not eligible to be included in this study:

* Subjects with other malignant tumors, excluding skin basal cell carcinoma and carcinoma in situ
* Presence of severe or uncontrollable systemic diseases, including uncontrollable hypertension or active bleeding tendency
* Patients judged by the investigator to be unsuitable for participation in the trial, or those with factors that may affect the patient's compliance with the protocol
* Toxicity caused by previous treatment has not recovered to normal state or is grade 1 according to NCI-CTCAE 5.0
* Allergic to or with metabolic disorders to the drugs in this protocol
* Pregnant or lactating women, or women with pregnancy plans during the study period and within 6 months after the last administration
* Patients participating in other clinical studies simultaneously

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2027-10-27 (Estimated); Study Completion 2027-10-27 (Estimated)

PRIMARY OUTCOMES:
Intracranial Overall Response Rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Intracranial overall response rate (iORR) is defined as the proportion of patients whose best overall response is either complete response (CR) or partial response (PR), as per local review and according to RANO-LM.

SECONDARY OUTCOMES:
Intracranial Progression Free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Intracranial progression-free survival (iPFS) is defined as the time from the date of randomization to the date of the first documented progression, as per local review and according to RANO-LM or death due to any cause.
Progression Free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Progression-free survival (PFS) is defined as the time from the date of randomization to the date of the first documented progression as per local review and according to RECIST 1.1 or death due to any cause.
Overall Survival | From date of randomization until the date of death from any cause, assessed up to 100 months
  Overall survival is defined as the time from the date of randomization to the date of death due to any cause
frequency/severity of adverse events, lab abnormalities | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial People's Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code